CLINICAL TRIAL: NCT01707576
Title: SCREENING OF ADOLESCENT MENTAL SUFFERING CONSULTANT TO EMERGENCIES, MANAGEMENT AND Later MONITORING
Brief Title: Screening of Adolescent Mental Suffering
Acronym: DESPERADOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry); Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P090103
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2010-01

CONDITIONS: Depression; Adolescent; Self-report Questionnaire
Keywords: Follow-Up Studies; Adolescent; Depressive Disorder, Major/diagnosis; Attempted/prevention & control; Self-report questionnaire; emmergency department; parental perception; Emergency
MeSH Terms: conditions — Depression; Depressive Disorder; Disease; Emergencies | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- screening of adolescent mental suffering. Management (Other): screening of adolescent mental suffering consultant to emergencies. Management and later monitoring
  Interventions: Behavioral: consultation 10 days later

INTERVENTIONS:
Behavioral: consultation 10 days later — new depression screening

SUMMARY:
The primary purpose is to estimate the prevalence of depression and subsyndromal states among adolescents 13 to 17 years consulting to hospital emergency rooms for any reason, for they are another way of tracking this suffering, as they host many troubled teens at once for health problems and accidents sometimes iterative, reflecting their risk behaviour.

Secondary purposes are to assess the feasibility and desirability of a post-emergency medical consultation for adolescents who scored high on a self-administered questionnaire, and to assess the impact of this approach by later monitoring.

DETAILED DESCRIPTION:
This is a multicenter longitudinal survey in three emergency centers in Ile-de-France, with 2 periods of daily collection and comprehensive three weeks spread over one year, followed by a remote evaluation.

The project is as follows:

Phase A :

- Evaluation of the prevalence: systematic execution of self-administered questionnaire by all adolescents consulting, night and day in each center.

Phase B :

* For adolescents whose outcome questionnaire exceed 4, a post-emergency consultation will be proposed within 15 days.
* Telephone survey, 12 months after the passage of emergency every teenager who completed self-administered questionnaire and presenting himself to the post-emergency consultation. This survey will aim to assess the psychological status of adolescents and the impact of any specific treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents over the age of 13 to 17 years when passing emergency whatever the reason for consultation (surgical or medical, including attempted suicide or psychological problem)

Exclusion Criteria:

* Young people not reading French.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 346 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Responses to Self-reported questionnaire on risk behaviors, somatic complaints by adolescents and parents | 10 months
  A self-questionnaire ADRS (Adolescent Depression Rating Scale) will be asked to all adolescents to complete. Also the other questions will be answered by them concenrning somatisations and risk behaviors. Parents respond in the same time a self questionnaire.

SECONDARY OUTCOMES:
Post-emergency consultation and reassessment of hetero-ADRS clinician questionnaire | 6 months
  Actual presence of adolescents suspected of depression at the post-emergency consultation and reassessment of their state using the hetero-ADRS-clinician questionnaire.

OTHER OUTCOMES:
Revaluation after one year | 6 months
  Revaluation after 1 year of the teenagers who come back to visit.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Stheneur, MD, Principal Investigator — Ambroise Paré University Hospital
Locations (1):
- Department of paediatric emergencies, Ambroise Paré universitary hospital, Boulogne-Billancourt, Île-de-France Region, France